CLINICAL TRIAL: NCT01161810
Title: Burn Patient Acuity Demographics, Scar Contractures and Rehabilitation Treatment Time Related to Patient Outcomes (ACT)
Brief Title: The Relationship of Rehabilitation Therapy Time To The Prevention of Burn Scar Contracture
Acronym: ACT
Status: Completed | Type: Observational
Sponsor: American Burn Association (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ABA-MCTG-0003; H-08-028 (Other Grant/Funding Number: US Army Institute of Surgical Research)
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Burns
Keywords: Burn; Rehabilitation
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post-Burn Rehabilitation: Patients with an acute burn injury who are admitted to the hospital with anticipated length of stay of 5 days or greater
  Interventions: Other: Routine post burn rehabilitation therapy

INTERVENTIONS:
Other: Routine post burn rehabilitation therapy — No testing outside of routine clinical rehabilitation will be performed

SUMMARY:
This project will develop a descriptive database of patient information and patient outcomes. This database will be used to determine the association of time spent in rehabilitation and patient outcomes, to relate patient acuity to burn scar contracture development and to establish minimal time requirement guidelines for various rehabilitation patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 year of age or older
* Admission for primary diagnosis of cutaneous burn injury
* Anticipated length of stay equal to/greater than five days
* >2% deep partial thickness burn OR hand burn (which may be less than 2% deep partial thickness burn)

Exclusion Criteria:

* Non-survivable burn as determined by the attending burn surgeon
* Electrical burn injury

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary diagnosis of acute burn injury
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2010-07; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Measure patient outcome in terms of time devoted to rehabilitation | At discharge
  Standard information that is recorded as part of daily routine in the rehabilitation treatment of patients with burn injury will be used as data to analyze patient outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Reginald L Richard, MS, PT, Principal Investigator — U.S. Army Institute of Surgical Research
Locations (14):
- United States (14):
  - Arizona Burn Center, Phoenix, Arizona
  - University of Califronia Irvine, Orange, California
  - University of California Davis, Regional Burn Center, Sacramento, California
  - Loyola University Health System, Maywood, Illinois
  - St. Joseph Regional Burn Center, Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Via Christi Regional Burn Center, Wichita, Kansas
  - Regions Hospital Burn Center, Saint Paul, Minnesota
  - St Elizabeth Regional Medical Center, Lincoln, Nebraska
  - NewYork-Presbyterian Weill Cornell Medical Center, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oregon Burn Center, Legacy Emanuel Hospital & Health Center, Portland, Oregon
  - U.S. army Institute of Surgical Research, Fort Sam Houston, Texas
  - University of Utah Health Services Center, Salt Lake City, Utah